CLINICAL TRIAL: NCT03307967
Title: Engaging Veterans Seeking Service-Connection Payments in Pain Treatment (PILOT)
Brief Title: Pilot of Pragmatic SBIRT Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); National Institute on Drug Abuse (NIDA) (NIH); US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2000022664_a; UG3AT009758 (NIH)
Record Dates: First submitted 2017-10-05; First posted 2017-10-12 (Actual); Results first posted 2022-05-16 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Substance Use Disorders; Pain
MeSH Terms: conditions — Substance-Related Disorders; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SBIRT-PM (Experimental): Screening, Brief Intervention and Referral to Treatment for Pain Management (SBIRT-PM) was developed to promote engagement in multi-modal non-pharmacological pain management among compensation-seeking Veterans with chronic pain. In SBIRT-PM, a clinician meets with the Veteran after the compensation examination to address the presenting MSD complaint. The clinician addresses Veterans' motivation for multi-modal pain care, and explains how pain can be managed using a variety of non-pharmacological pain management services. The clinician spells out how those services can be accessed at VA. Using permissive language about how pain is commonly self-medicated with substances, the clinician transitions to inquiries about use of prescription and non-prescription substances. The clinician then attempts to motivate Veterans to change their behavior if they are misusing substances. Thus, SBIRT-PM addresses the Veteran's presenting pain complaint first and nascent substance use subsequently.
  Interventions: Behavioral: SBIRT-PM

INTERVENTIONS:
Behavioral: SBIRT-PM — SBIRT-PM involves an initial telephone-delivered session followed by up to three calls to Veterans in a 12-week period to support Veteran engagement in multi-modal non-pharmacological pain care and to motivate those who misuse substances to change this problematic behavior. SBIRT-PM also includes coordination between the SBIRT-PM clinicians and the PACT nurse case manager after the initial session to support these patient outcomes.

SUMMARY:
Veterans seeking compensation for musculoskeletal (MSD) conditions often develop chronic pain and are at high risk for substance misuse. This study is designed to pilot test the Screening, Brief Intervention and Referral to Treatment for Pain Management (SBIRT-PM) intervention. SBIRT-PM is designed to reduce pain and reduce risky substance use among veterans applying for VA Benefits for a musculoskeletal condition, in part by helping Veterans get connected to comprehensive pain treatment. This pilot will involve a 2-year period to arrange for SBIRT Counselors at a single site to counsel Veterans throughout New England by phone with SBIRT-PM to test the acceptability and feasibility of the intervention.

DETAILED DESCRIPTION:
In 2015 alone, 97,223 new Veterans under age 35 began receiving compensation for injuries related to their military service. In total, there are 559,999 post-9/11 Veterans being compensated for back or neck conditions, and a partially overlapping 596,250 for limitation of flexion in joints. Veterans seeking compensation for musculoskeletal conditions often develop chronic pain and are at high risk for substance misuse. Early intervention is needed to arrest worsening pain and risky substance use, particularly among post-9/11 Veterans for whom engagement in non-pharmacological pain treatment has the potential to improve their overall quality of life and spare them the complications of opioid treatments. The service-connection application is an ideal point-of-contact for initiating early intervention treatments for these at-risk Veterans.

This study is designed to pilot test the Screening, Brief Intervention and Referral to Treatment for Pain Management (SBIRT-PM) intervention. SBIRT-PM is designed to reduce pain and reduce risky substance use among veterans applying for VA Benefits for a musculoskeletal condition, in part by helping Veterans get connected to comprehensive pain treatment. This pilot will involve a 2-year period to arrange for SBIRT Counselors at a single site to counsel Veterans throughout New England by phone with SBIRT-PM to test the acceptability and feasibility of the intervention.

During the two-years pilot trial, the team will prepare SBIRT-PM for implementation by establishing communication (Relational Coordination is the theoretical framework) between the "hub" where the SBIRT-PM clinician is sited and the "spoke" sites, establishing study-related procedures, and piloting the intervention at each of the eight VA medical centers in New England.

ELIGIBILITY:
Inclusion Criteria:

* Post-9/11 Veteran applying for MSD-related compensation, as ascertained from filed claim,
* Reports pain ≥4 on the pain Numerical Rating Scale (threshold for moderately severe pain);
* Availability of a landline or cellular telephone for SBIRT-PM.

Exclusion Criteria:

* Reports inability to participate during the study enrollment call
* Received three or more non-pharmacological pain treatment modalities (as previously categorized within the last 12 weeks from VA.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2019-06-17 (Actual); Study Completion 2019-06-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Rosen, MD, Principal Investigator — Yale University/ VA Connecticut Healthcare System; Steve Martino, PhD, Principal Investigator — Yale University/ VA Connecticut Healthcare System
Locations (2):
- United States (2):
  - Yale University, New Haven, Connecticut
  - VA Connecticut Healthcare System (VACHS), West Haven, Connecticut

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sellinger JJ, Martino S, Lazar C, Mattocks K, Rando K, Serowik K, Ablondi K, Fenton B, Gilstad-Hayden K, Brummett B, Holtzheimer PE, Higgins D, Reznik TE, Semiatin AM, Stapley T, Ngo T, Rosen MI. The acceptability and feasibility of screening, brief intervention, and referral to treatment for pain management among new England veterans with chronic pain: A pilot study. Pain Pract. 2022 Jan;22(1):28-38. doi: 10.1111/papr.13023. Epub 2021 Jun 26. PMID 33934499
- [Result] Rosen MI, Martino S, Sellinger J, Lazar CM, Fenton BT, Mattocks K. Access to Pain Care From Compensation Clinics: A Relational Coordination Perspective. Fed Pract. 2020 Jul;37(7):336-342. PMID 32908339

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Veterans in catchment area of New England VA Medical Centers applying for C&P disability benefits for a back, neck, knee, or shoulder condition
Period: Overall Study
Arm/Group | SBIRT-PM
Started | 40
Completed | 36
Not Completed | 4
Not completed — Lost to Follow-up | 4

BASELINE CHARACTERISTICS:
Arm/Group | SBIRT-PM
Number analyzed (Participants) | 40
Age, Continuous [Mean (Full Range); unit: years] | 40.2 [20 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 34
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 30
  Black | 3
  Other | 5
  Unknown | 2
  Hispanic | 6
Region of Enrollment [Number; unit: participants]
  United States | 40
Military Branch [Count of Participants; unit: Participants]
  Army | 18
  Marines | 5
  Navy | 7
  Airforce | 5
  Coast Guard | 2
  Army/Airforce | 2
  Army/Marines | 1

OUTCOME MEASURES:

1. Primary Outcome: Non-Pharm Pain Treatment Modalities Received
Description: A self-reported measure developed by the Pain Management Collaboaratory (PMC3). Questionnaire asks about the use of 13 different non-pharmacological pain treatments over the past 3 months. Below we present the mean number of non-pharmacological pain treatments received at baseline and then at week 12.
Time Frame: Baseline, Week 12
Measure: Mean (Standard Deviation); unit: non-pharm pain treatments
Arm/Group | SBIRT-PM
Number analyzed (Participants) | 36
non-pharm pain treatments
  # non-pharm pain treatments at Baseline | .93 (1.0)
  # non-pharm pain treatments at week 12 | 1.3 (1.3)

2. Primary Outcome: Substance Use
Description: Measured by the Alcohol, Smoking and Substance Involvement Screening Test (ASSIST). This self-reported assessment asks about the use of 10 classes of substances used over the preceding 3 months. In the below table, we present the number of participants that endorsed having used the indicated substance at baseline and week 12.
Time Frame: Baseline, week 12
Measure: Number; unit: participants
Arm/Group | SBIRT-PM
Number analyzed (Participants) | 36
participants
  Baseline : Alcohol | 13
  Baseline : Nicotine | 16
  Baseline : Other Drugs | 7
  Baseline : Alcohol or drugs | 27
  Week 12 : Alcohol | 6
  Week 12 : Nicotine | 15
  Week 12 : Other Drugs | 8
  Week 12 : Alcohol or drugs | 22

3. Primary Outcome: Change in Pain Severity
Description: Measured by the pain severity subscale of the Brief Pain Inventory (BPI). The BPI is a validated instrument to assess chronic non-cancer pain. The pain severity subscale consists of 4 items (worst pain, least pain, average pain, current pain) rated in the past 24 hours on a 0-10 scale- higher scores indicate higher pain severity. The four items are averaged to get a score. Below we present the mean, within-person change in pain severity from baseline to week 12. Minimally clinically important difference would be a 30% reduction in pain severity.
Time Frame: Baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: within-person change in score on a scale
Arm/Group | SBIRT-PM
Number analyzed (Participants) | 36
within-person change in score on a scale | -.41 (1.3)
Statistical Analysis 1: Comparison: SBIRT-PM; Test type: Other; p = .07, Wilcoxon (Mann-Whitney); Wilcoxon Signed Rank Sum

4. Primary Outcome: Change in Pain Interference
Description: Measured by the pain interference subscale of the Brief Pain Inventory (BPI). The BPI is a validated instrument to assess chronic non-cancer pain. The pain interference subscale consists of 7 items rated in the past 24 hours on a 0-10 scale- higher scores indicate higher interference from pain. The 7 items are averaged to get a score. Below we present the mean, within-person change in pain intensity from baseline to week 12. Minimally clinically important difference would be a 1 point reduction in pain intensity.
Time Frame: Baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: within-person change on a scale
Arm/Group | SBIRT-PM
Number analyzed (Participants) | 36
within-person change on a scale | .08 (1.6)
Statistical Analysis 1: Comparison: SBIRT-PM; Test type: Other; p = .98, Wilcoxon (Mann-Whitney); Wilcoxon Signed Rank Sum Test

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: An adverse event (AE) is any untoward medical occurrence in a subject during participation in the research study. Veterans with MSD have a high frequency of medical and psychiatric difficulties. Therefore, changes in medication regimen, the presence of medication side effects and symptom exacerbations are not untoward and do not constitute adverse events.
Arm/Group | SBIRT-PM
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 8/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SBIRT-PM (N=40)
Suicidal ideation (Psychiatric disorders) | 8 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-03-16): https://cdn.clinicaltrials.gov/large-docs/67/NCT03307967/Prot_SAP_000.pdf
  • Informed Consent Form (2020-05-12): https://cdn.clinicaltrials.gov/large-docs/67/NCT03307967/ICF_001.pdf